CLINICAL TRIAL: NCT02319772
Title: A Phase 1 Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BCX4430 Administered Via Intramuscular Injection (IM) in Healthy Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BCX4430
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCX4430-101; DMID 14-0030 (Other: NIAID/ Division of Microbiology and Infectious Diseases)
Record Dates: First submitted 2014-12-11; First posted 2014-12-18 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Filovirus Infections; Ebola Virus Infection
Keywords: Healthy volunteers; Ebola virus; Filovirus
MeSH Terms: conditions — Filoviridae Infections; Hemorrhagic Fever, Ebola | interventions — galidesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCX4430 (Experimental): BCX4430 administered as an IM injection
  Interventions: Drug: BCX4430
- Placebo (Placebo Comparator): Matched placebo administered as an IM injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCX4430
  Arms: BCX4430
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a 2-part, first-in-human dose-ranging study to evaluate the safety, tolerability and pharmacokinetics of escalating doses of BCX4430 administered via intramuscular (IM) injection in healthy subjects. In part 1, subjects will receive a single dose of BCX4430; in part 2 subjects will receive BCX4430 for 7 days.

DETAILED DESCRIPTION:
Part 1 of the study will evaluate the safety, tolerability and pharmacokinetics of single, ascending doses of BCX4430 versus placebo in healthy subjects. Up to 6 ascending dose cohorts will be enrolled in a sequential manner. Eight subjects will be treated with a single dose of study drug per dose cohort: 6 subjects per cohort will receive BCX4430, and 2 subjects per cohort will receive matching placebo.

Part 2 of the study will be initiated following review of all available data from Part 1 by an independent Safety Monitoring Committee

Part 2 of the study will evaluate the safety, tolerability, and pharmacokinetics of 7 days of daily dosing with BCX4430 versus placebo in healthy subjects. Up to 4 ascending dose cohorts will be treated in a sequential manner. Ten subjects will be treated with study drug per dose cohort (8 subjects will receive BCX4430 and 2 subjects will receive placebo per cohort). The planned doses and dosing regimens for each of the Part 2 cohorts will be determined based upon data collected during Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥ 50 kg (110 lbs) and ≤ 100 kg (220 lbs)
2. Body mass index (BMI) of 19-32 kg/m2
3. Willing to abstain from alcohol consumption for a period of 2 days prior to and during the study
4. Sexually active women of child bearing potential and sexually active men must utilize 2 highly effective contraceptive methods
5. Abstain from caffeinated beverages
6. Normal vital signs at rest
7. Ability to provide written informed consent

Exclusion Criteria:

1. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
2. Participation in a clinical research study within the previous 90 days
3. Any medical condition or medical history that, in the opinion of the investigator or sponsor, would interfere with the subject's ability to participate in the study or increase the risk of participation for that subject
4. Any screening laboratory test with an abnormal result that is grade 1 (mild) or greater
5. Abnormal ECG (defined as any screening or baseline QTc>450 msec, PR > 200 msec, or ventricular and/or atrial premature contractions that are more frequent than occasional, and/or as couplets or higher in grouping
6. An abnormal cardiovascular exam including a confirmed elevated blood pressure at screening (systolic greater than 140, diastolic greater than 90) after 5 minutes of supine rest, tachycardia >100 bpm after 5 minutes of supine rest
7. Family or personal history of sudden death or QT prolongation
8. Use of prescription, over-the-counter (OTC) medications or herbal supplements, with the exception of acetaminophen and non-oral hormonal contraception, for a period of 7 days prior to and during the study
9. Inadequate muscle mass to receive IM injections
10. History of alcohol or drug abuse within the previous year, or current evidence of substance dependence or abuse
11. Current smokers or history of smoking within the last 12 months
12. Serious adverse reaction or serious hypersensitivity to any drug
13. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
14. Donation or loss of greater than 400 mL of blood within the previous 3 months
15. Positive serology for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) type 1
16. Pregnant or nursing females
17. Male subjects with pregnant female partners

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety, measured by the frequency and severity of adverse events, laboratory abnormalities and other safety parameters following single (Part 1) and multiple (Part 2) doses of BCX4430 | Part 1: 7 days. Part 2: 14 days
  Evaluation of the incidence and severity of adverse events, laboratory abnormalities, ECG findings, vital sign changes, injection site and physical examination findings

SECONDARY OUTCOMES:
Plasma exposure of BCX4430, determined by the concentration time profile and PK parameters following single (Part 1) and multiple (Part 2) doses of BCX4430 | Part 1: 7 days. Part 2: 14 days
The urinary elimination of BCX4430, determined by the concentration of drug following single (Part 1) and multiple (Part 2) doses of BCX4430 | Part 1: 7 days. Part 2: 14 days

OTHER OUTCOMES:
The levels of BCX6870, the triphosphate metabolite of BCX4430, in peripheral blood mononuclear cells following single (Part 1) and multiple (Part 2) doses of BCX4430 | Part 1: 7 days. Part 2: 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jo Collier, MBChB, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Ruddington, United Kingdom

REFERENCES:
- [Derived] Mathis A, Collins D, Dobo S, Walling DM, Sheridan WP, Taylor R. Pharmacokinetics and Safety of the Nucleoside Analog Antiviral Drug Galidesivir Administered to Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2022 Apr;11(4):467-474. doi: 10.1002/cpdd.1037. Epub 2022 Feb 19. PMID 35182042